CLINICAL TRIAL: NCT04393493
Title: The Effect in Renal Function on Patients With Type 1 Cardiorenal Syndrome Treated With Two Strategies of Furosemide. A Randomized Controled Trial
Brief Title: The Effect in Renal Function on Patients With Type 1 Cardiorenal Syndrome Treated With Two Strategies of Furosemide.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Jonathan Samuel Chavez Iñiguez, MD, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112/17
Record Dates: First submitted 2017-08-22; First posted 2020-05-19 (Actual); Results first posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-08

CONDITIONS: Cardiorenal Syndrome
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — Chlorthalidone; Spironolactone

STUDY DESIGN:
Intervention Model Description: Its a randomized, controlled, phase II, 2-arm, double-blind clinical trial
Who Masked: Participant, Investigator
Masking Description: Double-blind clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP A (Experimental): Furosemide 80 mg every 24 hrs (morning) intravenously every 24 hrs for 4 consecutive days, additionally:
  * Day 1 furosemide 100mg / day infused with 100cc of Hartmann solution
  * Day 2 Furosemide 200mg / day infused with 100cc of Hartmann solution
  * Day 3 Furosemide 300mg / day infused with 100cc of Hartmann solution
  * Day 4 Furosemide 400mg / day infused with 100cc of Hartmann solution
  Interventions: Drug: Furosemide intravenous solution
- GROUP B (Experimental): Furosemide 80 mg every 24 hrs (morning) intravenously every 24 hrs for 4 consecutive days, additionally:
  * Day 1 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
  * Day 2 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
  * Day 3 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
  * Day 3 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
  Interventions: Drug: Furosemide intravenous solution; Drug: Chlortalidone; Drug: Spironolactone

INTERVENTIONS:
Drug: Furosemide intravenous solution — Administrated as an 80 mg intravenous bolus every 24 hours in both arms and then as a continuous infusion dosed according to the experimental arm.
Drug: Chlortalidone — One 50 mg pill administrated every 24 hours in group B
  Arms: GROUP B
Drug: Spironolactone — One 50 mg pill administrated every 24 hours in group B
  Arms: GROUP B

SUMMARY:
In double-blind clinical trial, determine renal recovery with two different furosemide strategies in patients with type 1 cardiorenal syndrome.

DETAILED DESCRIPTION:
In a patient with type 1 cardiorenal syndrome, we tried to compare two Furosemide strategies: both with a morning bolus, and randomized in two groups:

Group A: Furosemide 80 mg every 24 hrs (morning) intravenously every 24 hrs for 4 consecutive days, additionally:

* Day 1 furosemide 100mg / day infused with 100cc of Hartmann solution
* Day 2 Furosemide 200mg / day infused with 100cc of Hartmann solution
* Day 3 Furosemide 300mg / day infused with 100cc of Hartmann solution
* Day 4 Furosemide 400mg / day infused with 100cc of Hartmann solution

Group B: Furosemide 80 mg every 24 hrs (morning) intravenously every 24 hrs for 4 consecutive days, additionally:

* Day 1 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
* Day 2 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
* Day 3 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
* Day 4 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.

ution + Chlortalidone 50mg VO every 24 hours + Spironolactone 25mg VO every 24 hrs.

With the primary objective of improving renal function measured by serum creatinine, as secondary objectives the efficacy in vascular decongestion and electrolyte alterations.

ELIGIBILITY:
Inclusion Criteria:

* Comply with both clinical diagnosis of acute kidney injury by serum creatinine according to the Kidney Disease Improving Global Outcomes (KDIGO) 2012 guidelines and acute decompensate heart failure as clinical assessed by the clinical team in charge.
* Have agreed and signed informed consent

Exclusion Criteria:

* Patient in chronic dialysis either peritoneal dialysis or hemodialysis.
* History of being a renal transplant recipient
* History of acute kidney injury according to the KDIGO 2012 guidelines and / or renal replacement therapy in the last 3 months
* Pregnancy
* Impossibility to administer medication by the oral route

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - HCG, Guadalajara, Jalisco
  - Hospital Civil de Guadalajara, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chavez-Iniguez JS, Ibarra-Estrada M, Sanchez-Villaseca S, Romero-Gonzalez G, Font-Yanez JJ, De la Torre-Quiroga A, de Quevedo AA, Romero-Munoz A, Maggiani-Aguilera P, Chavez-Alonso G, Gomez-Fregoso J, Garcia-Garcia G. The Effect in Renal Function and Vascular Decongestion in Type 1 Cardiorenal Syndrome Treated with Two Strategies of Diuretics, a Pilot Randomized Trial. BMC Nephrol. 2022 Jan 3;23(1):3. doi: 10.1186/s12882-021-02637-y. PMID 34979962

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We screened all consecutive patients admitted for acute decompensated heart failure (ADHF) and acute kidney injury (AKI) who were evaluated by the Nephrology service at the Hospital Civil de Guadalajara Fray Antonio Alcalde, an University Hospital, from July 2017 to February 2020.
Pre-assignment Details: Of 168 patients assessed for eligibility, 80 met inclusion criteria and were randomized to treatment
Groups:
- Stepped Furosemide: Furosemide 80 mg every 24 hrs (morning) intravenously every 24 hrs for 4 consecutive days, additionally continuous infused furosemide as follows:
  * Day 1 furosemide 100mg / day infused with 100cc of Hartmann solution
  * Day 2 Furosemide 200mg / day infused with 100cc of Hartmann solution
  * Day 3 Furosemide 300mg / day infused with 100cc of Hartmann solution
  * Day 4 Furosemide 400mg / day infused with 100cc of Hartmann solution
- Diuretics Combined: Furosemide 80 mg every 24 hrs (morning) intravenously every 24 hrs for 4 consecutive days, additionally:
  * Day 1 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg orally every 24 hours + Spironolactone 25mg orally every 24 hrs.
  * Day 2 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg orally every 24 hours + Spironolactone 25mg orally every 24 hrs.
  * Day 3 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg orally every 24 hours + Spironolactone 25mg orally every 24 hrs.
  * Day 4 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg orally every 24 hours + Spironolactone 25mg orally every 24 hrs.
Period: Follow up
Arm/Group | Stepped Furosemide | Diuretics Combined
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0
Period: First 4 Days of Intervention
Arm/Group | Stepped Furosemide | Diuretics Combined
Started | 40 | 40
Completed | 35 | 33
Not Completed | 5 | 7
Not completed — Early improvement | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Stepped Furosemide: Furosemide 80 mg every 24 hrs (morning) intravenously every 24 hrs for 4 consecutive days, additionally:
  * Day 1 furosemide 100mg / day infused with 100cc of Hartmann solution
  * Day 2 Furosemide 200mg / day infused with 100cc of Hartmann solution
  * Day 3 Furosemide 300mg / day infused with 100cc of Hartmann solution
  * Day 4 Furosemide 400mg / day infused with 100cc of Hartmann solution
- Diuretics Combined: Furosemide 80 mg every 24 hrs (morning) intravenously every 24 hrs for 4 consecutive days, additionally:
  * Day 1 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
  * Day 2 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
  * Day 3 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
  * Day 4 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg VO every 24 hours + Spironolactone 50mg VO every 24 hrs.
- Total: Total of all reporting groups
Arm/Group | Stepped Furosemide | Diuretics Combined | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (14.5) | 59 (14.6) | 59 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 40 | 80
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Diabetes [Count of Participants; unit: Participants] — Hospital medical record of diabetes diagnosis or current use of antidiabetic drugs Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 39 | 38 | 77
    (all) | 25 | 30 | 55
Hypertension [Count of Participants; unit: Participants] — Hospital medical record of hypertension diagnosis or current use of antihypertensive drugs Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 39 | 38 | 77
    (all) | 29 | 35 | 64
Baseline serum creatinine [Mean (Inter-Quartile Range); unit: mg/dl] — Recorded serum creatinine form at least 3 months ago and up to one year ago
  mg/dl | 3.1 [2.2 to 4.7] | 2.8 [2.1 to 4] | 2.9 [2.2 to 4.5]
Chronic kidney disease [Count of Participants; unit: Participants] — Medical record of chronic kidney disease or as defined by KDIGO guidelines. Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 39 | 38 | 77
    (all) | 16 | 18 | 34
Baseline estimated glomerular filtration rate [Mean (Inter-Quartile Range); unit: ml/min/1.73m^2] | 31 [18 to 40] | 28 [16 to 58] | 28 [18 to 49]
Acute myocardial infarction [Count of Participants; unit: Participants] — Diagnosis of acute myocardial infarction by the cardiology service at admission.
  Our Hospital uses troponin levels, electrocardiographic changes and coronary angiography Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 38 | 37 | 75
    (all) | 8 | 8 | 16
Chronic heart failure [Count of Participants; unit: Participants] — Medical record of chronic heart failure diagnosis or previous echocardiographic study showing reduced left ventricular ejection fraction (<40%) or diastolic disfunction (elevated filling pressures). Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 39 | 37 | 76
    (all) | 26 | 24 | 50
Hypothyroidism [Count of Participants; unit: Participants] — Medical record of hypothyroidism diagnosis or diagnosed at hospitalisation with thyroid stimulating hormone and free T4 measures. Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 37 | 38 | 75
    (all) | 6 | 2 | 8
Arrythmia [Count of Participants; unit: Participants] — Medical record of any type of arrythmia or diagnosed at admission. Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 39 | 38 | 77
    (all) | 5 | 6 | 11
Current smoker [Count of Participants; unit: Participants] — Patient self reported current smoking Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 39 | 38 | 77
    (all) | 16 | 20 | 36
Heart rate [Mean (Inter-Quartile Range); unit: beats per minute] | 87 [80 to 99] | 82 [70.5 to 94] | 85 [72 to 98]
Oxygen saturation [Mean (Inter-Quartile Range); unit: percentage] — Individual average of measurements of one day before intervention started. Measurements made with pulse oximeter
  percentage | 95 [92 to 96] | 94 [92 to 96] | 94 [92 to 96]
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Individual average of measurements of one day before intervention started. Measurements made with a manual aneroid sphygmomanometer
  mmHg | 126 (23) | 134 (22) | 130 (23)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Individual average of measurements of one day before intervention started. Measurements made with a manual aneroid sphygmomanometer
  mmHg | 74 (12) | 77 (14) | 75 (13)
Uric acid [Mean (Inter-Quartile Range); unit: mg/dl] — First measurement during hospitalisation or most recent previous levels from up to 3 months ago. Population: Patients without the information required to assess this variable where excluded from the calculation
  mg/dl
    number analyzed (Participants) | 17 | 14 | 31
    (all) | 8.5 [8.1 to 9.5] | 9.1 [8.1 to 11.4] | 8.6 [8.1 to 10.3]
Presence of proteinuria in dipstick urinalysis [Count of Participants; unit: Participants] — Measured with the first dipstick urinalysis during hospitalisation Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 30 | 29 | 59
    (all) | 20 | 18 | 38
Presence of hematuria in dipstick urinalysis [Count of Participants; unit: Participants] — Measured with the first dipstick urinalysis during hospitalisation Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 30 | 29 | 59
    (all) | 19 | 15 | 34
Serum brain natriuretic peptide [Mean (Standard Deviation); unit: ng/dl] — Brain natriuretic peptide measured at admission as part of evaluation of acute heart failure Population: Patients without the information required to assess this variable where excluded from the calculation
  ng/dl
    number analyzed (Participants) | 11 | 13 | 24
    (all) | 2501 (1669) | 2718 (1836) | 2631 (1713)
Serum copeptin [Mean (Inter-Quartile Range); unit: ng/dl] — Levels measured at first day of intervention Population: Patients without the information required to assess this variable where excluded from the calculation
  ng/dl
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 75 [29 to 207] | 72 [49 to 115] | 75 [48 to 169]
Use of antibiotics at admission [Count of Participants; unit: Participants] — Antibiotic prescription at admission or at some point during hospitalisation Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 38 | 37 | 75
    (all) | 23 | 26 | 49
Blood transfusion during hospitalisation [Count of Participants; unit: Participants] — Requirement of blood transfusion at admission or at some point during hospitalisation.
  The indication was assessed by the clinical team in charge Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 37 | 37 | 74
    (all) | 3 | 1 | 4
Use of vasopressor drugs [Count of Participants; unit: Participants] — Prescription of vasopressor drugs at admission or during hospitalisation. Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 37 | 37 | 74
    (all) | 3 | 2 | 5
Use of inotropic drugs [Count of Participants; unit: Participants] — Prescription of inotropic drugs at admission or during hospitalization
  . Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 37 | 37 | 74
    (all) | 1 | 1 | 2
24 hr urinary volume before intervention [Mean (Inter-Quartile Range); unit: ml/day] — 24 hour urine volume measured one day before intervention started. Measurement was made by a nurse and the urine recollection was made through an urine catheter bag
  ml/day | 1278.93 [800 to 1475] | 1235.38 [762 to 1400] | 1266.57 [775 to 1450]
Use of normal saline as reanimation fluid [Count of Participants; unit: Participants] — Prescription of intravenous normal saline as reanimation or hydration fluid at admission or during intervention
  Participants | 2 | 2 | 4
Use of Hartmann solution as reanimation fluid [Count of Participants; unit: Participants] — Prescription of intravenous Hartmann solution as reanimation or hydration fluid at admission or during intervention Population: Patients without the information required to assess this variable where excluded from the calculation
  Participants
    number analyzed (Participants) | 40 | 39 | 79
    (all) | 27 | 29 | 56
Previous use of diuretics [Count of Participants; unit: Participants] — Patient self report of previous use of any type of diuretic drug in the last 3 months
  Participants | 10 | 6 | 16
Admission to internal medicine service [Count of Participants; unit: Participants] — Patients admitted from emergency department by the internal medicine service
  Participants | 24 | 23 | 47
Admission to cardiology service [Count of Participants; unit: Participants] — Patients admitted from emergency department by the cardiology service
  Participants | 14 | 14 | 28
Admission to intensive care unit [Count of Participants; unit: Participants] — Patients admitted from emergency department by the intensive care unit service
  Participants | 0 | 1 | 1
Admission to surgical service [Count of Participants; unit: Participants] — Patients admitted from emergency department by a surgical service
  Participants | 1 | 1 | 2
Admission to other hospital service [Count of Participants; unit: Participants] — Admission to other speciality service than the previously specified
  Participants | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Renal Function Recovery Defined as a Return to Individual Baseline Serum Creatinine Values
Description: Comparing patient's baseline serum creatinine (previous serum creatinine of 3 months ago and up to a year ago) with creatinine measurements every 24 hours during intervention (4 days)
Time Frame: Up to 96 hours after intervention started
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
Participants | 8 | 5

2. Secondary Outcome: Change in 24 Hour Urine Output at 96 Hours After Intervention Started From 24 Hour Urine Output One Day Before Intervention Initiation)
Description: Urine output was collected through an urinary catheter and measured and registered by a nurse. The sum of these registrations from 7 am from one day to 7 am of the next day was considered the 24 hour urinary output
Time Frame: 96 hours after intervention started
Measure: Mean (Inter-Quartile Range); unit: ml
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
ml | 125 [-350 to 1312] | 200 [-625 to 363]

3. Secondary Outcome: Change in Serum Creatinine at Day One of Intervention From Serum Creatinine at 96 Hrs After Intervention Started
Description: Calculated as serum creatinine at day one minus serum creatinine at 96 hrs after intervention started
Time Frame: 96 hours after intervention started
Measure: Mean (Inter-Quartile Range); unit: mg/dl
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
mg/dl | 0.02 [-0.3 to 0.6] | 0.2 [-0.02 to 0.5]

4. Secondary Outcome: An Elevation of at Least 0.3 mg/dl of Serum Creatinine From Day One of Intervention Compared With Serum Creatinine at 96hrs After Intervention Started
Time Frame: 96 hours after intervention started
Population: Patients without serum creatinine measured at 96hrs were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 37 | 35
Participants | 20 | 24

5. Secondary Outcome: In Hospital Mortality Defined as Number of Dead Patients From Day One of Intervention and Before Discharge
Time Frame: From day one of intervention up to discharge, an average of 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
Participants | 4 | 4

6. Secondary Outcome: Mortality During Follow up Defined as Number of Dead Patients After Discharge
Time Frame: From day one after discharge up to an average of 161 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 36 | 36
Participants | 9 | 12

7. Secondary Outcome: Number of Patients With Dyspnea Improvement as Referred by the Patient or Reduction in Supplementary Oxygen Requirements at 96 Hours After Intervention Started
Description: Dyspnea improvement was referred by the patient as the clinician asked them "do you feel more or less difficult to breathe?" or if the liters per minute or the fraction of inspired supplementary oxygen necessary to maintain an oxygen saturation >90% were diminished
Time Frame: Up to 96 hours after intervention started
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
Participants | 27 | 27

8. Secondary Outcome: Number of Patients With Dyspnea Improvement as Referred by the Patient or Reduction in Supplementary Oxygen Requirements Before Day 3 of Intervention
Description: Dyspnea improvement was referred by the patient as the clinician asked them "do you feel more or less difficult to breathe?" or if the liters per minute or the fraction of inspired supplementary oxygen necessary maintain an oxygen saturation >90% were diminished
Time Frame: Up to 3 days after intervention started
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
Participants | 2 | 7

9. Secondary Outcome: Number of Days From the Beginning of the Intervention Until Patients Referred Dyspnea Improvement or a Reduction in Supplementary Oxygen Requirements Was Made.
Description: as for outcome 8
Time Frame: Up to 4 days after intervention started
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
days | 4 [3 to 4] | 4 [2.2 to 4]

10. Secondary Outcome: Number of Patients That Required Renal Replacement Therapy of Any Type During Intervention (4 Days).
Description: The requirement of renal replacement therapy was assessed by the nephrology team in charge
Time Frame: Up to 96 hours after intervention started
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 38 | 38
Participants | 7 | 6

11. Other Pre Specified Outcome: Change in Serum Copeptin Levels at Day One of Intervention From Serum Copeptin Levels Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum copeptin levels at day one minus serum copeptin levels measured at 96 hrs after intervention started
Time Frame: 96 hours after intervention started
Population: Patients without the copeptin measurements made at day one and/or at 96hrs were excluded from this analysis
Measure: Mean (Inter-Quartile Range); unit: ng/dl
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 22 | 23
ng/dl | 1.1 [-20 to 21] | -16 [-26 to 13]

12. Other Pre Specified Outcome: Change in Serum Brain Natriuretic Peptide Levels at Baseline From Serum Brain Natriuretic Peptide Levels at 96 Hours After Intervention Started
Description: Baseline levels were defined as the measurement at hospital admission. Calculated as serum brain natriuretic peptide levels at baseline minus serum brain natriuretic peptide levels at 96 hours after intervention started
Time Frame: 96 hours after intervention started
Population: Patients without baseline brain natriuretic peptide measurements and/or without measurements at 96hrs were excluded from this analysis
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 7 | 9
ng/dl | -1344 (1041) | -1378 (1904)

13. Other Pre Specified Outcome: Number of Patients That Achieved >30% Reduction in Brain Natriuretic Compared With Baseline Levels
Description: Baseline levels were defined as the measurement at hospital admission
Time Frame: Up to 96 hours after intervention started
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 7 | 9
Participants | 5 | 7

14. Other Pre Specified Outcome: Number of Patients Whose Interventions Were Stopped Because Clinical Improvement Was Achieved Before 96 Hours as Assessed by de Clinical Judgement of the Medical Team in Charge.
Description: Clinical improvement was referred as remission of symptoms with achievement of 24 hour urine output equal or greater than 3000 milliliters
Time Frame: From the beginning of intervention and before 96 hours after that
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
Participants | 5 | 7

15. Other Pre Specified Outcome: Change in Serum Urea Levels Measured at Day One of Intervention From Serum Urea Levels Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum urea levels at day one of intervention minus serum urea levels at 96 hrs after intervention started.
Time Frame: 96 hours after intervention started
Measure: Mean (Inter-Quartile Range); unit: mg/dl
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
mg/dl | 13 [-11 to 37] | 18 [-1 to 45]

16. Other Pre Specified Outcome: Change in Serum Sodium Levels Measured at Day One of Intervention From Serum Sodium Levels Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum sodium levels at day one of intervention minus serum sodium levels at 96 hrs after intervention started.
Time Frame: 96 hours after intervention started
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
mEq/L | -1.2 (4.7) | 0.2 (4.7)

17. Other Pre Specified Outcome: Change in Serum Potassium Levels Measured at Day One of Intervention From Serum Potassium Levels Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum potassium levels at day one of intervention minus serum potassium levels at 96 hrs after intervention started.
Time Frame: 96 hours after intervention started
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
mEq/L | -0.2 (0.9) | -0.4 (0.8)

18. Other Pre Specified Outcome: Change in Serum Chloride Levels Measured at Day One of Intervention From Serum Chloride Levels Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum chloride levels at day one of intervention minus serum chloride levels at 96 hrs after intervention started.
Time Frame: 96 hours after intervention started
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
mEq/L | -0.6 (6.4) | -0.4 (4.7)

19. Other Pre Specified Outcome: Change in Serum Magnesium Levels Measured at Day One of Intervention From Serum Magnesium Levels Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum magnesium levels at day one of intervention minus serum magnesium levels at 96 hrs after intervention started.
Time Frame: 96 hours after intervention started
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
mg/dl | 0.07 (0.16) | -0.04 (0.2)

20. Other Pre Specified Outcome: Change in Serum Calcium Levels Measured at Day One of Intervention From Serum Calcium Levels Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum calcium levels at day one of intervention minus serum calcium levels at 96 hrs after intervention started.
Time Frame: 96 hours after intervention started
Measure: Mean (Inter-Quartile Range); unit: mg/dl
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
mg/dl | 0.15 [-0.4 to 0.6] | -0.05 [-0.2 to 0.3]

21. Other Pre Specified Outcome: Change in Serum pH Value Measured at Day One of Intervention From Serum pH Value Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum pH value at day one of intervention minus serum pH value at 96 hrs after intervention started.
Time Frame: 96 hours after intervention started
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
units | 0.03 (0.07) | 0.02 (0.04)

22. Other Pre Specified Outcome: Change in Serum Bicarbonate Levels Measured at Day One of Intervention From Serum Bicarbonate Levels Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum bicarbonate levels at day one of intervention minus bicarbonate levels at 96 hrs after intervention started.
Time Frame: 96 hours after intervention started
Measure: Mean (Inter-Quartile Range); unit: mEq/L
Groups:
- Diuretics Combined: Furosemide 80 mg every 24 hrs (morning) intravenously every 24 hrs for 4 consecutive days, additionally:
  * Day 1 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg orally every 24 hours + Spironolactone 25mg orally every 24 hrs.
  * Day 2 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg orally every 24 hours + Spironolactone 50mg orally every 24 hrs.
  * Day 3 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg orally every 24 hours + Spironolactone 50 orally every 24 hrs.
  * Day 4 furosemide 100mg / day infused with 100cc of Hartmann solution + Chlortalidone 50mg orally every 24 hours + Spironolactone 50mg orally every 24 hrs.
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
mEq/L | 2.9 [0.3 to 5.5] | 3 [1.1 to 4.7]

23. Other Pre Specified Outcome: Change in Serum Partial Pressure of Carbon Dioxide Measured at Day One of Intervention From Serum Partial Pressure of Carbon Dioxide Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum partial pressure of carbon dioxide at day one of intervention minus serum partial pressure of carbon dioxide at 96 hrs after intervention started.
Time Frame: 96 hours after intervention started
Measure: Mean (Inter-Quartile Range); unit: mmHg
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
mmHg | 1 [-2 to 6.7] | 3 [-1.5 to 6]

24. Other Pre Specified Outcome: Change in Serum Lactate Levels Measured at Day One of Intervention From Serum Lactate Levels Measured at 96 Hrs After Intervention Started.
Description: Calculated as serum lactate levels at day one of intervention minus serum lactate levels at 96 hrs after intervention started.
Time Frame: 96 hours after intervention started
Measure: Mean (Inter-Quartile Range); unit: mmol/L
Arm/Group | Stepped Furosemide | Diuretics Combined
Number analyzed (Participants) | 40 | 40
mmol/L | 0 [-0.3 to 0.4] | 0.1 [-0.2 to 0.3]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed at hospitalisation and during follow-up which lasted an average of 182 days. Serious adverse events and other adverse events were assessed during the 4 days that the intervention lasted.
Description: We assessed serious adverse events and other adverse events through daily clinical evaluation by one member of the nephrology team in charge and daily laboratory testing for serum creatinine, urea, glucose, sodium, potassium, chlorine, calcium, phosphorous, arterial or venous blood gas, and complete blood count.
  All cause mortality during follow-up was assessed through monthly phone calls to patients and/or searching at Hospital electronic records.
Arm/Group | Stepped Furosemide | Diuretics Combined
All-Cause Mortality (participants affected / at risk) | 13/40 | 16/40
Serious Adverse Events (participants affected / at risk) | 4/40 | 1/40
Other Adverse Events (participants affected / at risk) | 36/40 | 35/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stepped Furosemide (N=40) | Diuretics Combined (N=40)
Hypotension (Vascular disorders) | 4 (4) | 1 (1) — Any systolic blood pressure < 90mmHg and/or mean arterial pressure <65 mmHg
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stepped Furosemide (N=40) | Diuretics Combined (N=40)
Hypokalemia (Renal and urinary disorders) | 8 (8) | 7 (7) — Any serum potassium < 3.5 mEq/L during the intervention (4 days)
Hyponatremia (Renal and urinary disorders) | 18 (18) | 18 (18) — Any serum sodium < 3.5 mEq/L during the intervention (4 days)
Metabolic alkalosis (Renal and urinary disorders) | 12 (12) | 12 (12) — Any venous or arterial blood gas bicarbonate levels >28 mEq/L during the intervention (4 days)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04393493/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04393493/SAP_001.pdf